CLINICAL TRIAL: NCT06955208
Title: Evaluation of Meningioma Mechanical Properties and Histological Features Using Three-Dimensional Magnetic Resonance Elastography
Brief Title: 3D MRE-Based Evaluation of Meningioma Mechanical Properties and Histological Features
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Professor, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022_meningioma
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Meningioma
Keywords: Magnetic resonance elastography; Meningioma; Stiffness; Adhesion; Neurosurgery
MeSH Terms: conditions — Meningioma; Tissue Adhesions | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRE-Guided Surgery Group (Experimental): Participants in this group will undergo preoperative three-dimensional magnetic resonance elastography (3D MRE) in addition to routine MRI. MRE will be used to quantify tumor stiffness and generate a three-dimensional adhesion map. These imaging findings will be provided to the neurosurgical team prior to surgery to assist in planning the surgical approach and anticipating tumor consistency and adhesiveness. Intraoperative outcomes such as resection time, blood loss, and dissection difficulty will be recorded and analyzed in relation to preoperative MRE parameters.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography; Procedure: Intraoperative Assessment and Recording

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography — Participants will undergo preoperative 3D MRE to quantify tumor stiffness and generate adhesion maps. MRE is performed as an adjunct to standard brain MRI, using 60 Hz vibration frequency and specialized elastogram processing software. The resulting stiffness and adhesion data are made available to the neurosurgical team for surgical planning.
  Other Names: MRE
Procedure: Intraoperative Assessment and Recording — During surgical resection, the neurosurgical team will systematically assess and record tumor stiffness, adhesion to surrounding structures, vascularity, resection time, and technical difficulty using a standardized intraoperative scale. These intraoperative findings will be compared to preoperative MRE parameters to evaluate the diagnostic and predictive value of MRE.

SUMMARY:
This prospective single-center study aims to evaluate the feasibility and clinical utility of three-dimensional magnetic resonance elastography (3D MRE) in assessing tumor stiffness and adhesion in patients with meningioma undergoing surgical resection. By correlating preoperative MRE-derived stiffness and adhesion maps with intraoperative findings and histopathological features, the study seeks to determine whether MRE can serve as a noninvasive imaging biomarker for surgical planning, risk stratification, and prediction of tumor behavior.

DETAILED DESCRIPTION:
Meningiomas are the most common primary intracranial tumors and are often surgically resectable. However, the intraoperative texture and adhesion of the tumor to surrounding structures vary widely and directly impact the surgical approach, difficulty, and outcomes. Current preoperative imaging lacks the ability to quantitatively assess biomechanical properties such as stiffness and adhesion, which are critical for neurosurgical planning.

This prospective clinical trial investigates the application of 3D magnetic resonance elastography (MRE) in characterizing the biomechanical properties of meningiomas. Specifically, it aims to quantify tumor stiffness and adhesion using MRE-derived shear modulus maps and correlate these measurements with intraoperative surgeon-assessed stiffness/adhesion scores and postoperative histopathology. The study will also assess the diagnostic performance of MRE in predicting challenging resections, high tumor adhesion, and histological subtypes.

Approximately 300 patients with radiologically confirmed meningioma scheduled for elective resection will be enrolled. Participants will undergo standard MRI and additional 3D MRE scanning. Intraoperative findings including tumor stiffness, adhesion, blood supply, and resection difficulty will be systematically recorded. Postoperative pathological analysis will include tumor grade and histological subtype. Statistical analyses will evaluate correlations, diagnostic accuracy, and potential prognostic value.

Findings from this study may support the use of 3D MRE as a valuable noninvasive tool in preoperative assessment of meningiomas, helping optimize surgical strategies, reduce complications, and inform treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing meningeoma resection surgery are eligible for inclusion in the study cohort.

Exclusion Criteria:

* Patients with metallic implants or foreign bodies in their bodies (pacemakers, artificial metallic heart valves, metal joints, metal implants, and those who can not remove dentures, insulin pumps, or contraceptive rings)
* Pregnant women in the first trimester (within three months)
* Patients with severe claustrophobia or anxiety
* Patients with severe fever
* Patients who can not tolerate MRE
* Patients with vascular malformations and aneurysms.
* Patients who do not sign an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Agreement Between MRE Stiffness and Intraoperative Tumor Consistency | Intraoperative (Day of Surgery)
  The primary outcome is the correlation between preoperative 3D MRE-derived shear stiffness values and intraoperative tumor consistency as assessed by the neurosurgeon using a standardized ordinal scale (1-5). Agreement will be evaluated using Spearman correlation and Bland-Altman analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD, Principal Investigator — Shengjing Hospital; Anhua Wu, MD, Principal Investigator — Shengjing Hospital; Wen Cheng, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes JD, Fattahi N, Van Gompel J, Arani A, Meyer F, Lanzino G, Link MJ, Ehman R, Huston J. Higher-Resolution Magnetic Resonance Elastography in Meningiomas to Determine Intratumoral Consistency. Neurosurgery. 2015 Oct;77(4):653-8; discussion 658-9. doi: 10.1227/NEU.0000000000000892. PMID 26197204
- [Background] Yin Z, Lu X, Cohen Cohen S, Sui Y, Manduca A, Van Gompel JJ, Ehman RL, Huston J 3rd. A new method for quantification and 3D visualization of brain tumor adhesion using slip interface imaging in patients with meningiomas. Eur Radiol. 2021 Aug;31(8):5554-5564. doi: 10.1007/s00330-021-07918-6. Epub 2021 Apr 14. PMID 33852045
- [Background] Yin Z, Hughes JD, Trzasko JD, Glaser KJ, Manduca A, Van Gompel J, Link MJ, Romano A, Ehman RL, Huston J 3rd. Slip interface imaging based on MR-elastography preoperatively predicts meningioma-brain adhesion. J Magn Reson Imaging. 2017 Oct;46(4):1007-1016. doi: 10.1002/jmri.25623. Epub 2017 Feb 14. PMID 28194925